CLINICAL TRIAL: NCT05979168
Title: Effectiveness and Adoption of the Structured mHealth Intervention for Improving Blood Pressure Control (TelTex4BP) Among Adults With Hypertension in Nepal: A Randomized Controlled Trial
Brief Title: Effectiveness and Adoption of the TelTex4BP Intervention Among Adults With Hypertension in Nepal
Acronym: TelTex4BP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Department of Public Health (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BLSCHP-2303
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Hypertension; Medication Adherence; Blood Pressure; Cardiovascular Diseases
Keywords: Mobile Intervention; Blood Pressure Control; Hypertension; Randomized Controlled Trial
MeSH Terms: conditions — Hypertension; Medication Adherence; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This study will use a two-arm parallel-group, individually randomized control trial design to test the effectiveness of a TelTex4BP intervention compared to standard care at one year among diagnosed patients of HTN.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Hypertensive patients with uncontrolled BP in the intervention group will receive mobile phone text messages in the Nepali language and accept the phone call from the trained research nurse on their given mobile. They will also get the opportunity to ask questions and clarification during the phone call. However, text messaging would be only one way.
  Interventions: Behavioral: Phone call and text Messages
- Control arm (No Intervention): The control arm will receive the usual routine maintenance. In Nepal, hypertensive patients usually receive a prescription of antihypertensive medicine and advise for follow-up as the standard care. In addition, a pamphlet containing information about hypertension and required behavior modifications will be provided to all study participants, including the control arm.

INTERVENTIONS:
Behavioral: Phone call and text Messages — The intervention consists of recommended lifestyle counselling (on a healthy diet, physical activity, smoking, alcohol intake, medication adherence and continuity of care). This counselling will be provided through the research nurse at baseline and for six months (tentative plan phone call once a month; frequency and duration will be finalized based on formative study) by calling on participants' given mobile numbers. In addition, text message reminders on the same topics will be delivered regularly (2-3 times a week) for six months. The counselling and message will focus on three domains of COM-B; capabilities needed, opportunities and practical tools, and motivation strategies informed by behaviour change techniques.
  Other Names: TelTex4BP
  Arms: Intervention arm

SUMMARY:
Despite evidence of preventing cardiovascular disease (CVD) risk through lifestyle changes, many patients with hypertension (HTN) do not comply with this and suffer from CVD and other complications. A previous study using a structured lifestyle intervention program has reported a 14% decrease in the 10-year risk of developing CVD at one year among hypertensive and diabetes patients. Low and Middle-Income countries (LMICs) struggle with a shortage of health workers to deliver such interventions. In this context, mobile phones can contribute to bridging this gap by incorporating them into the health system for health intervention delivery. There is a need to develop contextual mHealth intervention adapted to local needs and culture and test its effectiveness in LMIC settings like Nepal. Our previous small-scale pilot mHealth (text messages) study reported promising evidence in reducing blood pressure among hypertensive patients in the intervention arm [adjusted reduction in systolic blood pressure (BP) -6.50 (95% CI, -12.6; -0.33) and diastolic BP -4.60 (95% CI, -8.16; -1.04)], with a greater proportion achieving target BP (70% vs 48% in the control arm, p = 0.006)] and improving treatment compliance (p < 0.001) in Nepal. This finding supports the expansion to a large-scale trial of a structured mHealth intervention to see its long-term effectiveness and sustainability for patients with HTN to improve BP control and reduce CVD risk. Hence, this study aims to assess the effectiveness of a behavioural intervention through mHealth (telephone/mobile phone calls and text messages) informed by the RE-AIM framework for improving blood pressure control among patients with hypertension in a hospital (Manamohan Cardiothoracic Vascular and Transplant Center) of Kathmandu, Nepal.

DETAILED DESCRIPTION:
This study will be a hybrid type 2 effectiveness-implementation study using mixed methods, a parallel randomized controlled trial with a nested qualitative design. The intervention will be codesigned involving patients, their family members, and healthcare providers to incorporate their views, the local context and culture through a formative qualitative component informed by the COM-B model. A multi-component mHealth intervention will be delivered through text messages and phone calls (TelTex4BP) by nurses, focusing on behaviour changes (physical activity, healthy diet), medication adherence, a reminder for follow-up, smoking, and alcohol intake. The intervention will be delivered for six months, and follow-up will be carried out at the end of the intervention and six months later (at one year) to assess sustainability and long-term effectiveness. Clinical (blood pressure, 10-year risk of CVD), intermediate (medication adherence, change of dietary habits/physical activity), and implementational outcomes ( Reach, Adoption, Intervention fidelity and Maintenance) will be evaluated using the RE-AIM framework. If the intervention is proven effective, the study findings will be disseminated to promote scaling up to other similar settings.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension
* Currently receiving/prescribed blood pressure-lowering medication for more than three month
* With uncontrolled blood pressure (>140/90mm of Hg)
* Should have access to a mobile phone
* Able to read text messages ( by themselves/with the help of family)

Exclusion Criteria:

* Diagnosed with myocardial infarction, stroke, and kidney failure
* Severe mental illness, cognitive impairment
* Pregnant women or in the postpartum period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | baseline, 6 and 12 months
  Average of last of two measures of Blood pressure.

SECONDARY OUTCOMES:
Blood Pressure Control | Baseline, 6 and 12 months
  Measures of Systolic and diastolic BP
10 year risk of development of CVD | Baseline, 6 and 12 months
  Globo CVD risk calculator
Medication adherence | Baseline, 6 and 12 months
  Hill-Bone compliance to high blood pressure therapy scale will be use to measure adherence to antihypertensive therapy. This tool contains 14 items: nine items related to medication, three items on salt intake and two items on appointment keeping. Each item is scored on a response of 1-4. The total score of Hill Bone is 56 where a lower score indicates higher adherence to antihypertensive therapy.
Dietary habits (salt intake, fruits and vegetables intake) | Baseline, 6 and 12 months
  Dietary salt [9 items] based on the WHO STEPs survey
Physical activity | Baseline, 6 and 12 months
  Physical activity [17 items]based on the WHO STEPs survey

CONTACTS AND LOCATIONS:
Overall Officials: Buna Bhandari Bhattarai, PhD, Principal Investigator — Central Department of Public Health, Tribhuvan University Institue of Medicine Nepal
Locations (1):
- Central Department of Public Health, Kathmandu, Pradesh 3 (Bagmati), Nepal

IPD SHARING:
Plan to Share IPD: No